CLINICAL TRIAL: NCT04896632
Title: A Randomized, Participant- and Investigator-blinded, Placebo-controlled, Single Ascending Dose and Multiple Dose Study to Assess the Safety, Tolerability, and Pharmacokinetics of INE963 in Healthy Participants
Brief Title: Study of Safety, Tolerability, and Pharmacokinetics of INE963 in Healthy Participants
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor's decision.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: CINE963A02101
Record Dates: First submitted 2021-05-12; First posted 2021-05-21 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- INE963 (Experimental): Part A is a single ascending dose (SAD) study with 7 planned cohorts Part B is a multiple dose (MD) study with 2 planned cohort q24h x 3 day of either INE963 or placebo
  Interventions: Drug: INE 963
- Placebo group (Placebo Comparator): Part A is a single ascending dose (SAD) study with 7 planned cohorts Part B is a multiple dose (MD) study with 2 planned cohort q24h x 3 day of either INE963 or placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: INE 963 — Part A: Single ascending dose with 7 planned cohorts> Part B: multiple dose with 2 planned cohort q24x3 days
  Arms: INE963
Other: Placebo — Part A: single ascending dose with 7 planned cohorts. Part B: multiple dose with 2 planned q24x3 days.
  Arms: Placebo group

SUMMARY:
The purpose of this study is to assess the safety, tolerability, and pharmacokinetics of single ascending doses and multiple doses of INE963 given orally in healthy participants.

DETAILED DESCRIPTION:
This is a randomized, participant- and investigator-blinded, placebo-controlled, single ascending and multiple oral dose study in healthy participants. The study consisted of two parts:

* Part A was a single ascending dose (SAD) study with 6 planned cohorts: (A1, A2, A4, A5, A6 and A7) of 8 participants each and 1 cohort (A3) with 10 participants, as randomization ratio 4:1 was originally planned due to the food effect cohort. There was also an optional cohort of 8 subjects (A8).
* Part B was a multiple dose (MAD) study with 2 planned cohort of 9 participants (B1 and B2; randomization ratio 2:1). There was also an optional cohort of 9 subjects (B3).

Cohort B2 and Optional Cohorts A8 and B3 were not dosed since the study was terminated early as per joint decision between the Principal Investigator and the Sponsor. Importantly, the decision to terminate the study early was not taken as a consequence of any safety concerns seen with INE963 administration in healthy volunteers.

ELIGIBILITY:
Inclusion criteria:

1. Written informed consent must be obtained before any assessment is performed.
2. Healthy male and female participants 18 to 55 years of age inclusive, and in good health as determined by past medical history, physical examination, vital signs, electrocardiogram, and laboratory tests at screening.
3. At screening and baseline, vital signs (systolic and diastolic blood pressure and pulse rate) will be assessed in the supine position Supine vital signs should be within the following ranges:

   * oral body temperature between 35.0 - 37.5 °C
   * systolic blood pressure, 90 - 140 mm Hg
   * diastolic blood pressure, 50 - 90 mm Hg
   * pulse rate, 40 - 90 bpm If vital signs are outside these ranges, the investigator may obtain up to 2 additional readings so that a total of up to 3 consecutive assessments are made. At least the last reading must be within the ranges provided above in order for the participant to qualify.
4. Participants must weigh at least 50 kg at screening and baseline to participate in the study, and must have a body mass index (BMI) within the range of 18.0 - 32.0 kg/m2. BMI = Body weight (kg) / [Height (m)]2
5. Able to communicate well with the investigator, to understand and comply with the requirements of the study.

Exclusion criteria

1. History of hypersensitivity to any of the study treatments or excipients or to drugs of similar chemical classes
2. Significant illness which has not resolved within two (2) weeks prior to initial dosing.
3. Recent (within the last three years of screening) and/or recurrent history of autonomic dysfunction (e.g., recurrent episodes of fainting, palpitations, etc.).
4. Recent (within the last three years of screening) and/or recurrent history of acute or chronic bronchospastic disease (including asthma and chronic obstructive pulmonary disease, treated or not treated).
5. Known history or current clinically significant arrhythmias.
6. Known family history or known presence of long QT syndrome.
7. A history of clinically significant ECG abnormalities, or any of the following ECG abnormalities at screening and/or baseline:

   * PR > 220 msec
   * QRS complex > 120 msec
   * RR >1.5 seconds
   * QTcF > 450 msec (males)
   * QTcF > 460 msec (females)
8. History of immunodeficiency diseases, including a positive HIV test result.
9. Chronic infection with Hepatitis B (HBV) or Hepatitis C (HCV). A positive HBV surface antigen (HBsAg) test, excludes a participant. Participants with a positive HCV antibody test should have HCV RNA levels measured. Participants with positive (detectable) HCV RNA should be excluded.
10. History of malignancy of any organ system (other than localized basal cell carcinoma of the skin or in-situ cervical cancer), treated or untreated, within the past 5 years of screening, regardless of whether there is evidence of local recurrence or metastases.
11. Donation or loss of 450 mL or more of blood within eight weeks prior to initial dosing, or longer if required by local regulation.
12. Plasma donation (> 450 mL) within 8 weeks prior to first dosing.
13. Any clinically significant hematology parameters outside normal ranges at screening and/or baseline. Participants with neutrophils <1.5 x 109/L should be excluded.
14. Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism, or excretion of drugs, or which may jeopardize the participant in case of participation in the study. The Investigator should make this determination in consideration of the participant's medical history and/or clinical or laboratory evidence of any of the following at screening or baseline:

    * Inflammatory bowel disease, peptic ulcers, gastrointestinal including rectal bleeding;
    * Major gastrointestinal tract surgery such as gastrectomy, gastroenterostomy, or bowel resection;
    * Pancreatic injury or pancreatitis;
    * Liver disease or liver injury as indicated by abnormal liver function tests (as defined below). ALT (SGPT), AST (SGOT), GGT, alkaline phosphatase and serum bilirubin will be tested.
    * Any single parameter of ALT, AST, GGT, alkaline phosphatase or serum bilirubin must not exceed the upper limit of normal (ULN)
    * History or presence of impaired renal function as indicated by clinically significantly abnormal creatinine or BUN and/or urea values, or abnormal urinary constituents (e.g. albuminuria).
    * Evidence of urinary obstruction or difficulty in voiding at screening.
15. Use of any prescription drugs, herbal supplements, prescribed medicinal use of cannabis/marijuana, within four weeks prior to initial dosing, and/or over-the-counter (OTC) medication, dietary supplements (vitamins included) within two weeks prior to initial dosing. If needed, (i.e. an incidental and limited need) paracetamol/acetaminophen is acceptable, but must be documented in the Concomitant medications / Significant non-drug therapies page of the CRF.
16. Smokers (use of tobacco/nicotine products 1 week prior to screening). Urine cotinine levels will be measured during screening and at each baseline for all participants. Smokers will be defined as any participant who reports tobacco use and/or who has a urine cotinine ≥ 200 ng/mL.
17. History of drug abuse or unhealthy alcohol use# within the 12 months prior to dosing, or evidence of such abuse as indicated by the laboratory assays conducted during screening and at baseline. #Unhealthy alcohol use is defined as a history of, or current alcohol misuse/abuse, defined as " >21 units for males and >14 units for females in the same week."
18. History of recreational cannabis use within four weeks prior to dosing, or evidence of such use as indicated by the laboratory assays conducted during screening and baseline. This exclusion criterion applies even if cannabis use is legalized where the site is located. Any prescribed, medicinal use of cannabis is to be handled according to the prescription drug usage criteria defined above.
19. Pregnant or nursing (lactating) women.
20. Sexually active males unwilling to use a condom during intercourse while taking investigational drug and for 5 half-lives or 14 days after stopping investigational drug, whichever is longer. A condom is required for all sexually active male participants to prevent them from fathering a child AND to prevent delivery of the investigational drug via seminal fluid to their partner for 5 half-lives or 14 days after last dose, whichever is longer. In addition, male participants should not donate sperm for the time period specified above. Additionally, the female partners of male participants should also use an effective method of contraception.
21. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant. Women are considered post-menopausal or not of child-bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or total hysterectomy at least six weeks before screening. In the case of oophorectomy alone, only when the reproductive status of the women has been confirmed by follow-up hormone level assessment if she is considered not of child-bearing potential. Refer to Section 8.6.6 Pregnancy and Assessments of Fertility.
22. Use of other investigational drugs at the time of enrollment or within 90 days of first dose in this study, or within 5 half-lives of enrollment, or until the expected PD effect has returned to baseline, whichever is longer; or longer if required by local regulations.
23. Participants who do not have suitable veins for multiple venipuncture cannulation as assessed by the investigator of delegate at screening
24. Participants in the food effect cohort: history of cholecystectomy or gall stones
25. Presence or history of clinically significant allergy requiring treatment as judged by the investigator. Hay fever is allowed unless it is active.
26. Evidence of an active infection, including COVID-19
27. Participants who are immediate family members to other participants
28. Participants who have previously participated in another cohort for this study
29. Known or current history of hemoglobinopathies including sickle cell disease
30. Intake of grapefruit or grapefruit juice within 14 days prior to initial dosing. No grapefruit or grapefruit juice is allowed until 7 days following the last dose

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2021-05-13 (Actual); Primary Completion 2022-11-24 (Actual); Study Completion 2022-11-24 (Actual)

PRIMARY OUTCOMES:
Number of Subjects with Significant Clinical Safety Labs, reporting SAEs and AEs and ECG findings | Dose escalation (21 days)
  Number of Subjects with Significant Clinical Safety Labs, reporting SAEs and AEs and ECG findings, as judged by investigator at each dose escalation review meetings

SECONDARY OUTCOMES:
INE963 pharmacokinetic parameters AUC in SAD Part | Day 1, 2, 3, 4, 6, 8, 9, 12 and 16
  INE963 pharmacokinetic parameters (AUC) in SAD Part at specified timepoints
INE963 pharmacokinetic parameters Tmax in SAD Part | Day 1, 2, 3, 4, 6, 8, 9, 12 and 16
  INE963 pharmacokinetic parameters in SAD Part (Tmax) at the specific timepoints
INE963 pharmacokinetic parameters Cmax in SAD Part | Day 1, 2, 3, 4, 6, 8, 9, 12 and 16
  INE963 pharmacokinetic parameters (Cmax) in SAD Part at specified timepoints
INE963 pharmacokinetic parameters Vz/F in SAD Part | Day 1, 2, 3, 4, 6, 8, 9, 12 and 16
  INE963 pharmacokinetic parameters in SAD Part (Vz/F) at the specific timepoints
INE963 pharmacokinetic parameters T1/2 in SAD Part | Day 1, 2, 3, 4, 6, 8, 9, 12 and 16
  INE963 pharmacokinetic parameters in SAD Part (T1/2) at the specific timepoints
INE963 pharmacokinetic parameters in MAD Part (AUC) | Day 1, 2, 3, 4, 6, 8, 10, 11, 14 and Day 18
  INE963 pharmacokinetic parameters in MAD Part (AUC) measured at specific timepoints
INE963 pharmacokinetic parameters in MAD Part (Cmax) | Day 1, 2, 3, 4, 6, 8, 10, 11, 14 and Day 18
  INE963 pharmacokinetic parameters in MAD Part (Cmax) measured at specific timepoints
INE963 pharmacokinetic parameters in MAD Part (Tmax) | Day 1, 2, 3, 4, 6, 8, 10, 11, 14 and Day 18
  INE963 pharmacokinetic parameters in MAD Part (Tmax) measured at specific timepoints
INE963 pharmacokinetic parameters in MAD Part (Vz/F) | Day 1, 2, 3, 4, 6, 8, 10, 11, 14 and Day 18
  INE963 pharmacokinetic parameters in MAD Part (Vz/F) measured at specific timepoints
INE963 pharmacokinetic parameters in MAD Part (T1/2) | Day 1, 2, 3, 4, 6, 8, 10, 11, 14 and Day 18
  INE963 pharmacokinetic parameters in MAD Part (T1/2) measured at specific timepoints
Baseline AAG concentration | Baseline
  Alpha-1- acid glycoprotein (AAG) level will be taken at baseline for Part A and Part b.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Mere Way, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No